CLINICAL TRIAL: NCT02774759
Title: Feasibility of the NEXT Steps Weight Loss Intervention +/- Resistance Training for Endometrial Cancer Survivors: Effect on Lean Mass & Biomarkers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015-1076; NCI-2016-00904 (Registry Identifier: NCI CTRP); 5T32CA101642 (NIH)
Record Dates: First submitted 2016-05-11; First posted 2016-05-17 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Malignant Neoplasms of Female Genital Organs
Keywords: Malignant neoplasms of female genital organs; Endometrial cancer survivors; Obese; Weight loss intervention; Resistance training; Aerobic exercise; Questionnaires; Surveys; Accelerometer; Fitness Test; Telephone Coaching; Video Chat Sessions
MeSH Terms: conditions — Obesity | interventions — Surveys and Questionnaires; Exercise Test; Resistance Training; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NEXT-Steps- Aerobic Exercise and Resistance Training (NS-ART) (Experimental): Participant wears an accelerometer for 7 days before baseline visit. Six questionnaires completed regarding quality of life and diet. Fitness test given covering various physical activities at baseline and at 6 month visit.
  Participants placed into an exercise plan focused on physical activity and resistance training. Physical activity guidelines workbook distributed along with activity monitor. Participants receive phone calls and text messages for support in reaching exercise and diet goals.
  Participants receive resistance bands to perform resistance exercises. Exercise handouts and an iPad mini with training videos used to video chat with a research team member.
  Questionnaires completed at 3 and 6 months regarding quality of life, diet, physical activity, etc.
  Interventions: Device: Accelerometer; Behavioral: Questionnaires; Behavioral: Fitness Test; Behavioral: Resistance Training; Behavioral: Telephone Coaching/Phone Calls; Behavioral: Video Chat Sessions
- NEXT-Steps- Aerobic Exercise (NS-A) (Experimental): Participant wears an accelerometer for 7 days before baseline visit. Six questionnaires completed regarding quality of life and diet. Fitness test given covering various physical activities at baseline and at 6 month visit.
  Participants placed into an exercise plan focused on physical activity only. Physical activity guidelines workbook distributed along with activity monitor. Participants receive phone calls and text messages for support in reaching exercise and diet goals.
  Questionnaires completed at 3 and 6 months regarding quality of life, diet, physical activity, etc.
  Interventions: Device: Accelerometer; Behavioral: Questionnaires; Behavioral: Fitness Test; Behavioral: Aerobic Exercise; Behavioral: Telephone Coaching/Phone Calls
- Standard Care Control Group (CG) (Active Comparator): Participant wears an accelerometer for 7 days before baseline visit. Six questionnaires completed regarding quality of life and diet. Fitness test given covering various physical activities at baseline and at 6 month visit.
  Participants receive standard of care consisting of phone calls asking about their health and self-help materials.
  Questionnaires completed at 3 and 6 months regarding quality of life, diet, physical activity, etc.
  Interventions: Device: Accelerometer; Behavioral: Questionnaires; Behavioral: Fitness Test; Behavioral: Telephone Coaching/Phone Calls

INTERVENTIONS:
Device: Accelerometer — Participant wears an accelerometer for 7 days before baseline visit to record activity levels, and again before their 6 month visit.
Behavioral: Questionnaires — Questionnaires completed at baseline regarding quality of life and diet.
  Questionnaires completed at 3 and 6 months regarding quality of life, diet, physical activity, etc.
  Other Names: Surveys
Behavioral: Fitness Test — Fitness test given covering various physical activities at baseline and at 6 month visit.
Behavioral: Resistance Training — Physical activity guidelines workbook distributed along with activity monitor. Participants receive resistance bands to perform resistance exercises. Exercise handouts and an iPad mini with training videos used to video chat with a research team member. Information from wireless scale and Fitbit sent to Fitbit website to monitor levels.
  Arms: NEXT-Steps- Aerobic Exercise and Resistance Training (NS-ART)
Behavioral: Aerobic Exercise — Participants placed into an exercise plan focused on physical activity only. Physical activity guidelines workbook distributed along with activity monitor.
  Arms: NEXT-Steps- Aerobic Exercise (NS-A)
Behavioral: Telephone Coaching/Phone Calls — Participants called 4 times during the first month, 2 times during the second month, and 1 time per month for the rest of the study. Participants also receive a follow-up call at the end of the study.
Behavioral: Video Chat Sessions — Video chatting between the research team and participants occurs 2 times per month during the first and third months, when new exercises are introduced. Video chatting offered monthly as needed by participants during months 2, 4, 5, and 6.
  Arms: NEXT-Steps- Aerobic Exercise and Resistance Training (NS-ART)

SUMMARY:
The goal of this research study is to learn if a home-based physical activity program is feasible and can help endometrial cancer survivors lose weight.

DETAILED DESCRIPTION:
Baseline Visit:

If participant is found to be eligible to take part in this study, an accelerometer will be mailed to them. An accelerometer is a small device that records participant's activity levels that participant wears on their waist during the day. Participant will wear this accelerometer for 7 days before their baseline visit. Participant will bring the accelerometer with them to the baseline visit.

Participant will also complete 8 questionnaires about their demographic information (such as their age, race, sex, and so on) / health and treatment history, current physical activity, quality of life, how well they function physically, sexual function, fatigue, body image, and safety as well as a brief survey about their exercise and nutrition preferences. It should take about 2 hours to complete the questionnaires and brief survey.

Participant will also complete 3 questionnaires online about what they ate in the last 24 hours. Two (2) will be completed during weekdays and the other on a weekend day. They should take about 45 minutes to complete. The link to the questionnaires will be emailed to participant.

At the baseline visit at MD Anderson:

* Participant's height, weight, blood pressure, and waist and hip circumferences will be measured.
* Blood (about 1½ tablespoons) will be drawn after participant fasts (has nothing to eat or drink but water) for 8 hours. These samples will be stored for future biomarker testing. Biomarkers will give information about inflammation, the breakdown of food into energy, and molecules released by fat cells. This information will help to see the changes in participant's metabolism and inflammation levels throughout the study.
* Participant will have a dual energy x-ray absorptiometry (DEXA) scan to check the amount of muscle in their body.
* Participant's fitness will be checked using a 6-minute walk test to see how far they can walk in 6 minutes. Participant will also see how many arm curls they can do in 30-seconds, how many times they can stand from a sitting position in 30-seconds, and how fast they can get out of a chair and walk 8 feet.

Study Groups:

After baseline, participant will be randomly assigned (as in the roll of the dice) to 1 of 3 study groups. Participant will have an equal chance of being in each group.

* If participant is in Group 1, they will have an exercise plan focused on physical activity and resistance training.
* If participant is in Group 2, they will have an exercise plan focused on physical activity only.
* If participant is in Group 3, they will receive the standard of care, which is phone calls asking about their health and self-help materials.

Study Procedures:

Both Groups 1 and 2:

* Participant will receive a portion control plate that they should use at least 1 time day to plan a meal.
* Participant will receive a personalized workbook with physical activity guidelines.
* Participant will be given a Fitbit (which measures their activity levels) and a wireless scale. The information from the scale and Fitbit will be sent to the Fitbit website so participant can monitor their activity levels. Participant can keep the Fitbit after the study is over, but they must return the scale.
* Participant will also be loaned an iPad mini if they do not own one. This can be used to video chat using FaceTime with the research team.
* Participant will be called 4 times during the first month, 2 times during the second month, and 1 time per month for the rest of the study. Participant will also receive a follow-up call at the end of the study. These calls can occur using the telephone or through video chat by using FaceTime on an iPad. The calls should take about 15-30 minutes. Participant will be asked for feedback on reaching goals, given tips for success, and helped to make plans that remove barriers to physical activity.
* Participant will receive around 7 text messages per week. Text messages will include feedback, support, and information about diet and exercise. Text messages will also ask participant to report how often they use their portion plate and how many servings of fruit and vegetables they ate during the day.
* Participant will be told to aerobic exercise (such as walking or swimming) for 30-60 minutes at least 5 days a week. The amount of exercise will slowly increase over the 6 months.

Group 1 only:

If participant is in Group 1, they will also use resistance exercise for 15-30 minutes at least 2 times a week. Participant will be given resistance bands, exercise handouts, and access to a video PDF containing training videos. Participant will use an iPad mini to video chat with a research team member twice during month 1 and once during month 3. Sessions will take between 30 and 60 minutes and will make sure participant is doing the exercises correctly and their questions are answered. Participant will need to return the loaned iPad mini after the study is over. Participant will be able to use their own iPad or iPad minis if they would like and will have electronic access to the necessary programs and videos.

Group 3:

If participant is in Group 3, they will be called 4 times during the first month, 2 times during the second month, and then 1 time a month for the remaining 4 months. Additionally, participant will receive a follow-up call at the end of the study. Participant will also receive self-help materials at 4 time points. Participants in this group will not receive a Fitbit, wifi scale, portion plate, or iPad mini.

Study Visits:

At 3 months, participant will be sent a link to 8 questionnaires about their physical activity, safety, satisfaction, quality of life, physical functioning, sexual function, body image and fatigue as well as brief survey. Participant will complete these online and it should take about 1½ hours to complete.

At 6 months participant will return to MD Anderson:

* Participant will complete 9 online questionnaires about their physical activity, diet, quality of life, satisfaction, safety, sexual function, fatigue, body image and ability to function physically. It will take about 3 hours to complete.
* Participant's height, weight, blood pressure and waist circumference will be measured.
* Blood (about 1½ tablespoons) will be drawn after participant fasts for 8 hours. These samples will be stored for biomarker testing as listed above.
* Participant will have a DEXA scan.
* Participant will repeat the fitness tests they did at their baseline visit which include a 6-minute walk test, 30-second arm curl, 30-second sit-to-stand test, and a test to see how fast they can get up from a chair and walk 8 feet.

The accelerometer will be mailed back to participant before their 6 month visit. Participant will be instructed to wear it again for 7 days, following the same instructions they were given for their first 7 days.

Length of Study:

Study participation will be over after participant completes the 6 month visit. Participant's study participation may be stopped early if they become injured, if they become ineligible (for example, if they need to have treatment), or if the research staff thinks it is in their best interest.

This is an investigational study.

Up to 75 participants will take part in the study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with Stage I-II endometrial cancer
2. Six to 36 months post treatment
3. Body mass index (BMI) 30-<45 kg/m2
4. Age of at least 18 years
5. Access to a telephone for coaching sessions and access to a computer, smartphone, or tablet for syncing Fitbit devices
6. Can speak and read English
7. Can provide informed consent
8. Willing to travel to MD Anderson's main campus for 2 visits (baseline and 6 months post-baseline)

Exclusion Criteria:

1. Unmanaged lymphedema
2. Medical contraindications to home-based exercise or low-fat, high fruit and vegetable diet
3. Functional limitations requiring a walker/scooter/wheelchair for daily activities
4. Recurrent disease
5. Vigorous exercise > or = 60 min/week or moderate exercise > or = 150 min/week. If a combination of moderate and vigorous exercise are preformed, the minutes of moderate exercise/week plus 2 x minutes of vigorous exercise/week > or = 150 min/week.
6. Resistance training on > or = 2 days/week accounting for more than 30 minutes of strength training per week
7. Enrollment in a structured weight loss program in the past 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-10-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Two Home-Based Weight Loss Interventions for Endometrial Cancer Survivors | 6 months
  Study considered feasible if consent rate is larger than 40%.
Feasibility of Two Home-Based Weight Loss Interventions for Endometrial Cancer Survivors | 6 Months
  Study considered feasible if retention rate is larger than 70%.
Feasibility of Two Home-Based Weight Loss Interventions for Endometrial Cancer Survivors | 6 months
  Study considered feasible if adherence in NEXT Steps- Aerobic exercise and Resistance Training (NS-ART) and NEXT Steps- Aerobic exercise (NS-A) is larger than 65%.
Feasibility of Two Home-Based Weight Loss Interventions for Endometrial Cancer Survivors | 6 months
  Study considered feasible if the mean overall satisfaction with the program is larger than 3.5 in a 5-level scale.

SECONDARY OUTCOMES:
Changes in Lean Body Mass | 6 months
  Changes in lean body mass measured by dual-energy x-ray absorptiometry (DXA).

CONTACTS AND LOCATIONS:
Overall Officials: Karen Basen-Engquist, PHD, BA, MPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org